CLINICAL TRIAL: NCT06392490
Title: Evaluation of the Effectiveness of a Technology-based Program Delivered by Peer-led and Adult Educators to Adolescents Diagnosed With Asthma
Brief Title: The Effectiveness of Peer-education Programs for Adolescents Diagnosed With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Emine Güneş Şan, Phd candidate, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-Gazi-SBE-E.896440
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Asthma; Adolescent Behavior; Self Efficacy; Peer Support and Chronic Disease
Keywords: Asthma; Adolescent; Information; Education; Pediatric; Randomized controlled trial; Quality of life; Self-management; Technology; Internet; Nursing
MeSH Terms: conditions — Asthma; Adolescent Behavior; Chronic Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer Group (Other): -The experimental group that will apply the technology-based psychosocial program from peers
  Interventions: Other: Technology Based Asthma Program
- Adult Group (Other): -The group that will apply the technology-based psychosocial program from adult
  Interventions: Other: Technology Based Asthma Program
- Control Group (No Intervention): Control group that will no apply the technology-based psychosocial program

INTERVENTIONS:
Other: Technology Based Asthma Program — Evaluate the impact of peer-led and adult-based technology-based education on the quality of life, asthma control, asthma knowledge and self-efficacy in adolescents diagnosed with asthma.
  Arms: Adult Group; Peer Group

SUMMARY:
The research was planned in a randomized controlled trial to evaluate the effect of technology-based education provided by peers and adults to children diagnosed with asthma in the 14-17 age group. The study will be conducted in two phases. The initial phase will assess the efficacy of the training provided to peer mentors. The subsequent phase will examine the impact of peer-led and adult-delivered technology-based education on quality of life, asthma control, asthma knowledge, and self-efficacy in adolescents diagnosed with asthma. The required institutional permission and ethics committee approval was received. The study group of the study will consist of 48 adolescents (intervention group 1 [n=16], intervention group 2 [n=16], and control group [n=16]). Data will be collected by using the descriptive features form, the Adolescent Asthma Self-Efficiacy Questionaire, the Asthma Quality of Life Scale for Children, the Asthma Control Test, the Asthma Knowledge Test.The data will be analyzed using the SPSS 27 program.

DETAILED DESCRIPTION:
Asthma is the most common chronic disease in children. Although asthma often occurs in childhood, it can occur at any age. The incidence and prevalence of asthma is higher in children. On average, 5-10% of the world's population has an individual diagnosed with asthma, and one-third of these individuals are under the age of 18. In the United States of America (USA), approximately 6 million children between the ages of 0-17 are diagnosed with asthma. It has been reported that adolescents are at high risk for poor asthma outcomes, and death rates from asthma are twice as high in the 11-17 age group than in the 0-10 age group.

Peer relationships and peer support are of particular importance for children with chronic illnesses. Adolescents diagnosed with asthma value support from their peers. Adolescents tend to seek guidance from people with similar characteristics, and the opinions of individuals with similar characteristics are more valuable than those of individuals who do not have similar characteristics. Being with an adolescent diagnosed with asthma can improve the adolescent's sense of support and sense of normalcy. It is crucial to create an environment where adolescents diagnosed with asthma can interact with other adolescents diagnosed with asthma, thereby facilitating the formation of a support network.The research was planned in a randomized controlled trial to evaluate the effect of technology-based education provided by peers and adults to children diagnosed with asthma in the 14-17 age group. The study group of the study will consist of 48 adolescents (intervention group 1 [n=16], intervention group 2 [n=16], and control group [n=16]). The technology-based program will be applied to adolescents for 4-6 weeks through modules on the website. At the end of the study, it will apply website modules to the adolescents in the control group. The research is based on the Bandura's Self-Efficacy Theory.

ELIGIBILITY:
Inclusion Criteria:

* the ages of 14 and 17 who have been diagnosed with asthma at least three months prior
* who do not have any other medical diagnoses of chronic disease.
* who must own and be able to use a smartphone, reliable home internet access, and a computer.
* who must be proficient in Turkish and not be in the active attack period.
* who must not have experienced a stressful event that could affect their quality of life in the last three months, such as an acute illness, the birth of a new sibling, or the death of a family member.

Exclusion Criteria:

* who are unwilling or unable to continue the research
* who fail to participate in the internet-based application on two or more occasions

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Adolescent Asthma Self-Efficacy Questionnaire | Change from Baseline level to 3 months (change is being assessed)
  The scale is applied to adolescents aged 12-18 with a diagnosis of asthma. Scale items are scored from 0 to 100. The responses to the scale items are added and then divided by 27 to obtain the total average score (0-100). Subscale items are added in the same way and divided by the number of items in each subscale. A higher score indicates higher self-efficacy.
Asthma Quality of Life Scale for Children | Change from Baseline level to 3 months (change is being assessed)
  The instrument was developed to assess the physical, mental and social disorders of children diagnosed with asthma in the 7-17 age group. The scores range from 23 to 161. The items on the scale are evaluated using a 7-point Likert scale. A high score indicates a high quality of life, while a low score indicates a low quality of life.
Asthma Control Test | Change from Baseline level to 3 months (change is being assessed)
  The Asthma Control Test (ACT) is a five-item instrument designed to assess asthma control. The ACT scores range from 5 to 25, with a score of 5 indicating poor asthma control and a score of 25 indicating complete control of asthma. A score below 19 is generally used to indicate uncontrolled asthma.
Asthma knowledge test | Change from Baseline level to 3 months (change is being assessed)
  This form will be created by researchers in accordance with the existing literature. It will be used to evaluate information about asthma symptoms, triggers and treatment. The form will be created in a 3-point Likert type as "True", "False" and "I don't know". In the form, each correct answer will receive "1 point", while incorrect answers and those marked "I don't know" will receive "0 points". A high total score obtained from this form will indicate a high level of knowledge about asthma.

CONTACTS AND LOCATIONS:
Locations (1):
- Emine Gunes San, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data (IPD) available to other researchers